CLINICAL TRIAL: NCT06985342
Title: A Prospective, Open-Label Study Examining the Use of Rimegepant ODT 75 mg or Zavegepant Nasal Spray 10 mg for Acute Treatment of Migraine in the Emergency Department Setting
Brief Title: Acute Migraine Treatment in the ED With Gepants
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jonathan Schimmel, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-01677
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Migraine Headaches
Keywords: Migraine; Emergency Department; Gepants; CGRP antagonists; Rimegepant; Zavegepant
MeSH Terms: conditions — Migraine Disorders; Emergencies | interventions — rimegepant sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rimegepant (Experimental): Participants in this arm will receive a single dose of rimegepant 75 mg orally disintegrating tablet (ODT) for acute migraine treatment during an Emergency Department (ED) encounter.
  Interventions: Drug: Rimegepant
- Zavegepant (Experimental): Participants in this arm will receive a single dose of zavegepant 10 mg nasal spray for acute migraine treatment during an Emergency Department (ED) encounter.
  Interventions: Drug: Zavegepant

INTERVENTIONS:
Drug: Rimegepant — Rimegepant 75 mg orally disintegrating tablet (ODT), administered as a single dose
  Arms: Rimegepant
Drug: Zavegepant — Zavegepant 10 mg nasal spray, administered as a single dose
  Arms: Zavegepant

SUMMARY:
This study evaluates the effectiveness of rimegepant 75 mg orally disintegrating tablet (ODT) single-dose or zavegepant 10 mg nasal spray single-dose as acute migraine treatments during Emergency Department (ED) encounters. Although these two calcitonin gene-related peptide receptors (CGRP) receptor antagonists are FDA-approved for the indication of acute migraine treatment, past studies have been limited to the outpatient setting. If these medications are effective in the Emergency Department, their delivery methods alone may have advantages over intravenous medications commonly used for acute migraine in EDs, including quicker time to treatment delivery, faster pain relief, and reduced ED length of stay. This investigation is a pilot study to examine rimegepant and zavegepant in an ED, to gain insight on effectiveness in this setting.

This study will administer rimegepant 75 mg ODT single-dose or zavegepant 10 mg nasal spray single-dose as acute migraine treatments to 100 patients in the Emergency Department. It is a single center, open-label, non-controlled 2-group clinical trial (allocated 1:1 to rimegepant or zavegepant via pseudo-random assignment). The study will enroll adults in the ED meeting ICHD-3 criteria for migraine or probable migraine, with or without aura.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Capacity to provide informed consent (without a Legally Authorized Representative)
* Prior migraine diagnosis (clinical or self-reported)
* Emergency Department presentation for a headache fulfilling International Classification of Headache Disorders (ICHD-3) criteria for migraine with typical aura or without aura, or criteria for probable migraine with typical aura or without aura. Duration of migraines should be ≥ 1 year. It is acceptable if current headache duration is >72 hours. Must have been headache free for >48 hours prior to current attack.
* Willingness to participate in post-discharge telephone or electronic follow-up assessments

Exclusion Criteria:

* Suspected secondary headache due to another cause, or primary headache disorder other than migraine or probable migraine
* Prior healthcare encounter for headache within 7 days
* Use of analgesics or abortive headache medications within 2 hours of consent
* Use of intranasal decongestant within 12 hours of consent
* Use of the following drug/food categories with potential for drug interactions within 7 days or 5 half-lives, whichever is longer: 1) CYP3A strong or moderate inducers, 2) CYP3A4 strong inhibitors, 3) P-glycoprotein (P-gp) inhibitors, 4) OATP1B3 transporter potent inhibitors/inducers, 5) NTCP transporter potent inhibitors/inducers
* History of cardiovascular disease, hypertension, or diabetes, recently diagnosed or currently uncontrolled or unstable
* History of stroke, peripheral vascular disease, or medically-diagnosed Raynaud's Phenomenon
* History of severe hepatic impairment, as assessed by the investigator or qualified delegate
* History of kidney disease stage 4 (creatinine clearance <30 mL/min or eGFR <35 mL/min/1.73 m2)
* History of nasal condition that may affect zavegepant administration, as assessed by the investigator or qualified delegate
* History of hypersensitivity reaction to rimegepant, zavegepant, or to any included inactive ingredients
* Lifetime use of CGRP-targeting acute or preventive migraine medications
* In custody of law enforcement
* Current pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with pain relief at 2 hours without rescue medication | 120 minutes (2 hours)
  Percentage of participants reporting pain as 'mild' or 'none' at 2 hours post-study drug administration, without rescue medication. Pain is categorized as none, mild, moderate, or severe.

SECONDARY OUTCOMES:
Percentage of participants with pain relief at 2 hours post treatment | 120 minutes (2 hours) post treatment
  Effectiveness of treatment measured as percentage of participants with pain relief achieving "mild" or "none" at 2 hours post-study drug administration. Pain is categorized as none, mild, moderate, or severe.
Percentage of participants with pain relief at 60 minutes post treatment | 60 minutes post treatment
  Effectiveness of treatment measured as percentage of participants with pain relief achieving "mild" or "none" at 60 minutes post-study drug administration. Pain is categorized as none, mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Schimmel, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan does not include sharing of patient-level data.